CLINICAL TRIAL: NCT05021393
Title: Impact of Clinical Pharmacist Intervention as a Part of the Multidisciplinary Team on Clinical Outcomes in Cancer Patients With Pain in Nepal: A Feasibility Pilot Randomized Controlled Trial (PharmCaP Trial)
Brief Title: Clinical Pharmacists' Intervention on Pain Management in Cancer Patients
Acronym: PharmCaP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University Malaysia (Other)
Responsible Party: Principal Investigator, Sunil Shrestha, Principal Investigator, Monash University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: PharmaCAP trial
Record Dates: First submitted 2021-08-17; First posted 2021-08-25 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Cancer; Cancer Pain
Keywords: cancer; cancer pain; clinical pharmacist; multidisciplinary team; pain intensity; quality of life
MeSH Terms: conditions — Neoplasms; Cancer Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive the services from a clinical pharmacist and the existing standard care available in the medical oncology ward.
  Interventions: Other: Clinical Pharmacist Intervention
- Control Group (No Intervention): The standard care includes the current existing care provided to patients in the hospital. In addition, it includes all the available medical and non-medical services except the service provided by the clinical pharmacist.

INTERVENTIONS:
Other: Clinical Pharmacist Intervention — Medication review, patient education, counseling, and corresponding written recommendation will be performed by clinical pharmacists for all randomized patients.
  Arms: Intervention Group

SUMMARY:
The study aims to evaluate the impact of clinical pharmacist intervention as a part of a multidisciplinary team to improve clinical outcomes of cancer patients with pain in comparison to standard care.

DETAILED DESCRIPTION:
For the intervention group, medication review, patient education, counseling, and recommendation will be performed by clinical pharmacists for all randomized patients. Patient education and counseling include giving education regarding drugs used in pain management, their adverse drug reactions. Medication review includes assessing the appropriateness of each of the regular medications based on laboratory findings, medication lists, consultation and discharge notes, procedures, and test results. Face-to-face interviews will be conducted with patients prior to the follow-up. Clinical pharmacists will assess drug use history used for pain management, identify drug-related problems, identify ADRs and provide drug therapy interventions through written pharmacist notes to physicians during the follow-up, based on the medication chart review and the above pharmaceutical assessments.

After the follow-up, the clinical pharmacist will educate on drug-related problems identified before the visit, reinforce physician's instruction, and encourage drug compliance using written patient educational leaflets. Telephone follow follow-up will be conducted 4 weeks after the visit. Patients randomized to the control group will attend the medical follow-up as usual and receive usual care. All patients will be followed up for 4 weeks post-intervention visits. Data collection will be conducted at baseline and 4 weeks after the pharmacist visit. The primary outcome of the study is pain intensity which will be measured at baseline (prior to physician visit), and at 4 weeks post-intervention follow-up.

Patients will be encouraged to keep in touch with the clinical pharmacist through various communication tools (including short messages, mobile phone contact, or Viber or WhatsApp). They will be also encouraged to request a consultation for any pain control issue at any time.

This prospective randomized controlled trial will be conducted in the cancer hospitals of Nepal.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 18 years old, diagnosed with cancer, and had self-reported cancer pain within a month prior to the study.
2. Patients be able to read and understand the Nepalese language or English language.
3. the patient is under standard analgesia treatments.
4. the patient was estimated to have over 2 months of survival time.
5. Access to a telephone or mobile phone or internet
6. The patients must understand the study process and evaluation, agree to participate in this trial, and sign the informed.

Exclusion Criteria:

1. Patients who self-reported to have severe cognitive impairments.
2. Patients who are unable to complete pain assessment.
3. Participating in any other investigational therapies or other study protocols that may impact pain intensity are the primary outcomes of this study.
4. History of drug abuse, history of drug addiction, or severe alcoholism.
5. Opioid allergy.
6. Critically ill patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 4 weeks
  NRS was used to assess pain intensity. The responses were given using an eleven-point numeric rating scale (NRS) scored 0-10, where 0 = best outcome/does not interfere/no pain/complete pain relief and 10 = worst outcome/completely interferes/most pain/no pain relief.

SECONDARY OUTCOMES:
Change in Quality of life | 4 weeks
  EORTC QLQ-C30 (Version 3) uses for questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 (Version 3) uses for questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, the raw score has to be calculated with mean values. An afterward linear transformation is performed to be comparable. More points are considered to have a better outcome.
Edmonton Symptom Assessment System (revised version) | 4 weeks
  The revised Edmonton Symptom Assessment System (ESAS-r) is designed to assess 10 common symptoms: pain, tiredness, drowsiness, nausea, lack of appetite, shortness of breath, depression, anxiety, well-being, and constipation.
  The patient circles the most appropriate number to indicate where the symptom is between "0" and "10". "0" is the minimum value, which means there is no change and it is a better outcome for the patient. "10" is the maximum value, which means that the symptom level is the highest, which is a worse outcome for the patient.
Adverse Drug Reaction | 4 weeks
  Adverse events will be assessed throughout the study according the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) Version 4.0. Number of subjects who experienced an adverse event in this study is presented.
Medication Adherence | 4 weeks
  Medication Adherence Report Scale-5 (MARS-5): Changes in self-reported adherence using the MARS-5 at 4 weeks post-baseline. The MARS-5 assesses adherence to treatment.
  The MARS-5 assesses a patient's typical medication adherence through 5 questions (eg, "I forget to take my medication"; "I alter the dose of my medication"), using a 5-level response format (1-always, 2-often, 3-sometimes, 4-rarely, and 5-never).
Hospital Anxiety and Depression | 4 weeks
  Hospital Anxiety and Depression Scale (HADS): The Hospital Anxiety and Depression Scale (HADS), a self-assessment scale, was developed to detect states of depression, anxiety and emotional distress amongst patients who were being treated for a variety of clinical problems.
  The HADS includes 14 items assessing anxiety (7-item) and depression (7-item), which are rated on a 4-point Likert-type (from 0 to 3). The scores in each subscale are computed by summing the corresponding items, with maximum scores of 21 for each subscale. A score of 0-7 is considered as normal, 8-10 as a borderline case, and 11-21 as a case (anxiety or depression)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Shrestha, Principal Investigator — Monash University Malaysia
Locations (2):
- Nepal (2):
  - Kathmandu Cancer Center, Bhaktapur, Bagmati
  - Civil Service Hospital, Kathmandu, Bagmati

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shrestha S, Blebil AQ, Teoh SL, Sapkota S, Kc B, Paudyal V, Gan SH. Clinical pharmacists' intervention on pain management in cancer patients (PharmaCAP trial): study protocol for a randomized controlled trial. J Pharm Policy Pract. 2023 Jan 24;16(1):14. doi: 10.1186/s40545-022-00505-0. PMID 36694232
- [Derived] Shrestha S, Sapkota S, Teoh SL, Kc B, Paudyal V, Lee SWH, Gan SH. Clinical pharmacist interventions on pain management in cancer patients (PharmaCAP) in low resource settings: a multicenter feasibility-pilot randomized controlled trial. Support Care Cancer. 2024 Nov 27;32(12):828. doi: 10.1007/s00520-024-08989-z. PMID 39601933